CLINICAL TRIAL: NCT00287521
Title: A Study of Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-68
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open; angle; glaucoma; ocular; hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — Latanoprost

ARMS (4):
- AL-37807 Suspension (Experimental)
  Interventions: Drug: AL-37807 Ophthalmic Suspension, 1.0%
- Xalatan (Active Comparator)
  Interventions: Drug: Latanoprost, 0.005% (Xalatan)
- AL-37807 Vehicle (Placebo Comparator)
  Interventions: Other: AL-37807 Vehicle
- Timolol Maleate (Experimental)
  Interventions: Drug: Timolol Maleate Ophthalmic Gel Forming Solution, 0.5%

INTERVENTIONS:
Drug: AL-37807 Ophthalmic Suspension, 1.0% — One drop in the study eye(s) once daily for 28 days
  Arms: AL-37807 Suspension
Drug: Latanoprost, 0.005% (Xalatan) — One drop in the study eye(s) once daily for 28 days
  Other Names: XALATAN
  Arms: Xalatan
Other: AL-37807 Vehicle — One drop in the study eye(s) once daily for 28 days
  Arms: AL-37807 Vehicle
Drug: Timolol Maleate Ophthalmic Gel Forming Solution, 0.5% — One drop in the study eye(s) once daily for 28 days
  Arms: Timolol Maleate

SUMMARY:
The purpose of this study is to determine whether a glaucoma therapy is safe and effective in treating patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma (with ot without pseudoexfoliation or pigment dispersion component) or ocular hypertension
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 18
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Mean intra-ocular pressure (IOP) change at Day 28 from baseline (Day 0) | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- United States Investigative Sites in Texas and Other States, Fort Worth, Texas, United States